CLINICAL TRIAL: NCT02396537
Title: Efficacy of Topical Lidocaine to Decrease Discomfort With Intranasal Midazolam Administration: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Efficacy of Topical Lidocaine to Decrease Discomfort With Intranasal Midazolam Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Christopher Pruitt, Pediatric Emergency Medicine Faculty Advisor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: F130917005
Record Dates: First submitted 2015-03-11; First posted 2015-03-24 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Pain
Keywords: Children; Midazolam; Lidocaine; Intranasal
MeSH Terms: conditions — Pain | interventions — Lidocaine; Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Lidocaine (Experimental): Patient to receive 4% lidocaine intranasally prior to midazolam
  Interventions: Drug: Lidocaine; Drug: Midazolam
- Intranasal 0.9% saline (Placebo Comparator): Patient to receive 0.9% Saline intranasally prior to midazolam
  Interventions: Drug: Midazolam; Drug: 0.9% Saline

INTERVENTIONS:
Drug: Lidocaine — Administered intranasally prior to Midazolam administration.
  Other Names: Xylocaine
  Arms: Intranasal Lidocaine
Drug: Midazolam — Administered to all patients immediately after study drug (Lidocaine or Placebo) administered.
  Other Names: Versed
Drug: 0.9% Saline — Administered intranasally prior to Midazolam administration.
  Arms: Intranasal 0.9% saline

SUMMARY:
The purpose of this study was to establish whether premedication with topical lidocaine would reduce the pain associated with IN midazolam administration in children. The study was designed to be a double-blinded, randomized, placebo-controlled trial performed in an urban, academic pediatric emergency department.

DETAILED DESCRIPTION:
This was a double-blinded, randomized, placebo-controlled trial performed in an urban, academic pediatric emergency department with an annual census of 67,000 patients. Children 6-12 years old for whom IN midazolam was ordered were eligible for enrollment. Patients were randomly assigned an identical intranasal medication (4% Lidocaine or 0.9% saline). Patients were administered the study drug followed by IN midazolam. Patients then assigned a pain score for midazolam administration using the Wong-Baker FACES Pain Rating scale. The primary endpoint of pain score was analyzed with a two-tailed Mann-Whitney U test, with P < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-12
* Previously healthy
* Attending physician concludes that the patient would benefit from administration of an anxiolysis medication prior to a minor procedure

Exclusion Criteria:

* Moderate to severe asthma or other chronic lung disease
* Co-morbid conditions including cerebral palsy, developmental delay, or other chronic illness deemed by the Attending physician to be unsafe to receive anxiolysis with Versed.
* Any child presenting with a life-threatening condition.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, Principal Investigator — UAB Department of Pediatrics

REFERENCES:
- [Derived] Smith D, Cheek H, Denson B, Pruitt CM. Lidocaine Pretreatment Reduces the Discomfort of Intranasal Midazolam Administration: A Randomized, Double-blind, Placebo-controlled Trial. Acad Emerg Med. 2017 Feb;24(2):161-167. doi: 10.1111/acem.13115. Epub 2017 Jan 30. PMID 27739142

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Lidocaine | Intranasal 0.9% Saline
Started | 40 | 37
Completed | 40 | 36
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Lidocaine | Intranasal 0.9% Saline | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [7 to 10] | 9 [7 to 10] | 8 [7 to 10]
Gender [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 38 | 36 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 23 | 22 | 45
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: Discomfort With Intranasal Midazolam Administration
Description: subject self-reports pain with intranasal midazolam utilizing the Wong-Baker FACES Pain Scale. This scale is a well-established ordinal pain scale for pediatric patients. It is one score (no subscales), with a minimum score of 0 (signifying "No Hurt") and a maximum score of 10 ("Hurts Worst"). Values between include 2 ("Hurts Little Bit"), 4 ("Hurts Little More"), 6 ("Hurts Even More"), and 8 ("Hurts Whole Lot."). Children indicate one value/answer. Thus, a higher score indicates a worse outcome (more pain).
Time Frame: immediately after administration of intranasal midazolam
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Intranasal Lidocaine: Subjects were administered 4% lidocaine solution, 0.5 ml in each naris, 5 minutes prior to intranasal midazolam (intervention group).
- Intranasal 0.9% Saline: Subjects were administered 0.9% saline, 0.5 ml in each naris, 5 minutes prior to intranasal midazolam (placebo group).
Arm/Group | Intranasal Lidocaine | Intranasal 0.9% Saline
Number analyzed (Participants) | 40 | 36
units on a scale | 3 [0 to 6] | 8 [2 to 9]

ADVERSE EVENTS:
Time Frame: duration of study (8 months)
Arm/Group | Intranasal Lidocaine | Intranasal 0.9% Saline
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/37
Other Adverse Events (participants affected / at risk) | 0/40 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No